CLINICAL TRIAL: NCT03574675
Title: Acute Exposure of Simulated Hypoxia on Non-invasive Cardiac Output Assessments at Rest and During Exercise
Brief Title: Acute Exposure of Simulated Hypoxia on Cardiac Output
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2018-00455_A6
Record Dates: First submitted 2018-06-20; First posted 2018-07-02 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Pulmonary Hypertension
Keywords: simulated altitude; exercise; non-invasive cardiac output
MeSH Terms: conditions — Hypertension, Pulmonary; Motor Activity

STUDY DESIGN:
Intervention Model Description: Including a baseline assessment and assessments under simulated altitude and normoxia
Who Masked: Participant
Masking Description: The allocated gas mixture will not be disclosed to the patient since he will breath trough a facemask during both interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Order Sham/Hypoxia (Experimental): The participants will be consecutively exposed to shamed hypoxia (FiO2: 20.9%) equivalent to sea level and to simulated altitude (FiO2: 15.1%) equivalent to 2500m above sea level administered by an altitude simulator ("Altitrainer", SMTEC) with a facemask.
  Interventions: Device: Simulated Altitude (FiO2: 15.1); Device: Shamed Hypoxia (FiO2: 20.9)
- Order Hypoxia/Sham (Experimental): The participants will be consecutively exposed to hypoxia (FiO2: 15,1%) equivalent to 2500m above sea level and to shamed hypoxia (FiO2: 20.9%) equivalent to sea level administered by an altitude simulated ("Altitrainer", SMTEC) with a facemask.
  Interventions: Device: Simulated Altitude (FiO2: 15.1); Device: Shamed Hypoxia (FiO2: 20.9)

INTERVENTIONS:
Device: Simulated Altitude (FiO2: 15.1) — Inhalation of deoxygenated air through an altitude simulator ("Altitrainer") for approximately 1 hour given by a facemask.
Device: Shamed Hypoxia (FiO2: 20.9) — Inhalation of unmodified air through an altitude simulator ("Altitrainer") for approximately 1 hour given by a facemask.

SUMMARY:
Randomized crossover trial in patients with Pulmonary Hypertension (PAH, CTEPH) to assess the acute response to simulated altitude (FIO2: 15.1% = equivalent to 2500m above sea level) on non-invasive cardiac output assessments by Finapres® "NOVA" Technology at rest and under exercise.

DETAILED DESCRIPTION:
Low altitude baseline measurements will be performed in Zurich (470m asl) including Echocardiography, right heart catheterization, six-minute walk test (6MWT), pulmonary function test, clinical assessment and blood gas analysis at rest and under exercise.

Randomly assigned to the order of testing, the participants will be tested under simulated altitude (FiO2: 15.1% with the "AMC Altitrainer") and shamed altitude with the same device.

During the exposure to simulated altitude (FiO2: 15.1%) and shamed altitude of 1 hour each, the participants cardiac output non-invasively assessed will be measured throughout the whole intervention.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* PH diagnosed according to internation Guidelines: mean pulmonary artery pressure (mPAP) ≥ 25 mmHg along with a Pulmonary artery Wedge pressure (PAWP) ≤15 mmHg during right heart catheterization at the time of initial diagnosis
* PH class 1 (PAH) or 4 (CTEPH)
* Stable condition, on the same medication for > 4 weeks
* Patient live permanently at an altitude < 1000m asl.

Exclusion Criteria:

* Resting partial oxygen pressure (PaO2) ≤7.3 kiloPascal (kPA) corresponding to the requirement of long-term oxygen therapy > 16hour daily (nocturnal oxygen therapy alone is allowed)
* Severe daytime hypercapnia (pCO2 > 6.5 kPa)
* Susceptibility to high altitude related diseases (AMS, High Altitude Pulmonary Edema (HAPE), etc.) based on previous experienced discomfort at altitudes.
* Exposure to an altitude >1500m for ≥3 nights during the last 4 weeks before the study participation
* Residence > 1000m above sea level
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, neurological or orthopedic problems with walking disability
* Women who are pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Cardiac Output measured non-invasively | 1 hour
  Change in non-invasive assessed cardiac output measured with a finger cuff (Finapres) during the exposure to simulated altitude (FiO2: 15.1%) compared to normoxia

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Ulrich, MD, Principal Investigator — University of Zurich
Locations (1):
- Respiratory Clinic, University Hospital of Zurich, Zurich, Switzerland